CLINICAL TRIAL: NCT01142258
Title: Trazodone for the Treatment of Sleep Disorders in Alzheimer's Disease: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: Trazodone for Sleep Disorders in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Collaborators: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Einstein Francisco de Camargos, MD, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZD-001
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Sleep; Sleep Disorders; Insomnia; Alzheimer's Disease
Keywords: Sleep Disturbances; Alzheimer disease; Insomnia; Trazodone; Treatment
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Alzheimer Disease; Parasomnias | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trazodone (Experimental): Study group will receive trazodone 50mg
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): Inert pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — Trazodone tablets, 50 mg, 10pm (before bedtime) for 14 days.
  Arms: Trazodone
Drug: Placebo — Inactive or inert pill which will be used as a comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether trazodone is effective in the treatment of sleep disorders in Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Sleep disorders (SD) affects 35 to 50 percent of patients with AD. These disorders often make caring for patients at home very difficult. Trazodone is commonly prescribed drugs for SD in AD patients. There are no controlled studies in this sample of patients for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Fifty-five years of age or older;
* Diagnosis of probable Alzheimer's disease by National Institute of Neurological and Communicative Disorders and Stroke/the Alzheimer's Disease and Related Disorders Association criteria;
* Hachinski Ischemia Scale score less than 5
* Mini-Mental State Examination score of O to 26
* Actigraph evidence of a mean time immobile of less than 7 hours per night based on at least 7 nights of complete actigraph data collected over a single week;
* For-week history of sleep disorder behaviors, occurring at least once weekly, as reported by the caregiver using the Neuropsychiatric Inventory (NPI) Nighttime Behavior scale;
* Sleep disturbance observed was not present before the diagnosis of AD;
* Other co-morbidities, especially delirium, depression, chronic pain and medication use may be present, but do not cooperate in the primary symptoms;
* Computed tomography or magnetic resonance imaging since the onset of memory problems showing no more than 1 lacunar infarct in a nonstrategic area and no clinical events suggestive of stroke or other intracranial disease or normal;
* Stable medications for 4 weeks prior to the screening visit;
* Having a mobile upper extremity to which to attach an actigraph;
* Residing with a responsible spouse, family member, or professional caregiver who is present during the night and would agree to assume the role of the principal caregiver for the 3-week protocol;
* Ability to ingest oral medication and participate in all scheduled evaluations

Exclusion Criteria:

* Sleep disturbance associated with an acute illness, delirium or psychiatric disease;
* Clinically significant movement disorder, such as akinesia, that would affect actigraphic differentiation of sleep and wakefulness
* Severe agitation;
* Unstable medical condition;
* Discontinuation of psychotropic or sleep medications within 2 weeks of the screening visit;
* Patient unwilling to maintain caffeine abstinence after 2:00 PM for the duration of the protocol;
* Patient unwilling to comply with the maximum limit of 2 alcoholic drinks per day, and only 1 alcoholic drink after 6:00 PM for the duration of the protocol;
* Prior use of trazodone for the treatment of sleep disturbances;
* Caregiver deemed too unreliable to supervise the wearing of the actigraph, to administer trazodone the proper time, to maintain tbe sleep diary, or to bring the patient to the scheduled visits;

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Nighttime Total Sleep Time | Baseline, 14 days follow-up

SECONDARY OUTCOMES:
Change from Baseline in Nighttime Wake After Sleep Onset | Baseline, 14 days follow-up
Change from Baseline in Nighttime Number Of Awakenings | Baseline, 14 days follow-up
Change from Baseline in Daytime Total Sleep Time | Baseline, 14 days follow-up
Change from Baseline in Number of Daytime Naps | Baseline, 14 days follow-up
change in cognitive function (as measured by the Mini-Mental State Examination) | Baseline, 14 days follow-up
Change in activities of daily living (The index of ADL - Katz) | Baseline, 14 days follow-up
Change of baseline in behavioral variables (BAHAVE-AD scale) | Baseline, 14 days follow-up
Proportion of subjects who gained at least 30 minutes in total nighttime sleep | Baseline, 14 days follow-up
Change from Baseline in Clinical Dementia Rating | Baseline, 14 days follow-up
Change from Baseline in cognitive function (Digit Symbol Substitution Test) | Baseline, 14 days follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Einstein F Camargos, MD, MsC, Principal Investigator — Brasilia University - Brasilia's University Hospital - Geriatric Medical Centre
Locations (1):
- Geriatric Medical Centre, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- [Derived] Camargos EF, Louzada LL, Quintas JL, Naves JO, Louzada FM, Nobrega OT. Trazodone improves sleep parameters in Alzheimer disease patients: a randomized, double-blind, and placebo-controlled study. Am J Geriatr Psychiatry. 2014 Dec;22(12):1565-74. doi: 10.1016/j.jagp.2013.12.174. Epub 2014 Jan 4. PMID 24495406